CLINICAL TRIAL: NCT05229718
Title: Understanding and Optimizing Care for Young Adults With Type 1 and Type 2 Diabetes Mellitus Transitioning to the Adult Diabetes Care Setting
Brief Title: Understanding and Optimizing Care for Young Adults With Type 1 and Type 2 Diabetes Mellitus Transitioning to Adult Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Deborah Wexler, MD, Clinical Director MGH Diabetes Center, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021P002431
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-05

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: Young Adults; Emerging Adults; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care Model (Active Comparator): Patients enrolled in this arm will receive diabetes care per usual care at the Massachusetts General Hospital (MGH) Diabetes Center.
  Interventions: Other: Usual Care Model
- Diabetes Collaborative Care Model for Young Adults (Active Comparator): Patients enrolled in this arm will receive diabetes care per the diabetes collaborative care model for young adults.
  Interventions: Other: Diabetes Collaborative Care Model for Young Adults

INTERVENTIONS:
Other: Diabetes Collaborative Care Model for Young Adults — We designed a diabetes collaborative care model for young adults that incorporates a mental health provider alongside a diabetes care provider during joint office visits to facilitate screening and treatment of psychosocial determinants of diabetes management. The Massachusetts General Hospital (MGH) Diabetes Center will be piloting this model with a multi-disciplinary team of diabetologists, nurse practitioners, diabetes nurse educators, and mental health provider. Patients scheduled to be seen in the diabetes collaborative care model will continue to follow in the diabetes collaborative care model, with follow up visits every 3-4 months. All patients will receive routine diabetes care with lab testing, medical interventions, therapies and referrals performed at the discretion of the patients' providers.
  Arms: Diabetes Collaborative Care Model for Young Adults
Other: Usual Care Model — Patients enrolled in this arm will receive routine diabetes care per usual care at the Massachusetts General Hospital (MGH) Diabetes Center, with lab testing, medical interventions, therapies and referrals performed at the discretion of the patients' providers. In the usual care model, behavioral/mental health and social work services are available on a referral basis and are not integrated into a patients' routine appointment. Screening and treatment of psychosocial determinants of diabetes management are at done at the discretion of the patients' provider. Frequency of follow up visits is at the discretion of the patients' provider.
  Arms: Usual Care Model

SUMMARY:
In this study, we will determine the feasibility of an innovative care model for young adults with diabetes and compare the primary and secondary outcomes in the innovative model to those in the usual care model for adult diabetes management at Massachusetts General Hospital (MGH) Diabetes Center.

DETAILED DESCRIPTION:
This study is a quasi-randomized mixed methods evaluation of the implementation of an innovative collaborative care model to assess whether it is feasible and improves indicators of diabetes and mental health, while exploring themes that will inform redesign of the care model to improve healthcare delivery to young adults with diabetes transitioning to the adult care setting. We will compare primary and secondary outcomes in this model to those in the usual care model for adult diabetes management at MGH Diabetes Center. Those who agree to the research study will be asked to complete a series of three survey questionnaires over the timeframe of the study. The electronic health records (EHRs) of these patients who agree to the research study will also be examined. All patients who successfully complete all 3 survey questionnaires will be eligible for a structured interview portion of the study to explore themes that will inform care model redesign.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes mellitus
* Between ages 18 and 30 years
* Any duration of diabetes
* Must self-manage diabetes
* A new patients at the Massachusetts General Hospital (MGH) Diabetes Center at 50 Staniford Street as of September 1, 2021.
* The patient does not have to be diagnosed with diabetes in youth or have been previously seen at MGH for Children (MGHfC) Pediatric Diabetes Clinic to be included

Exclusion Criteria:

* Patients with gestational diabetes, diabetes during pregnancy, MODY, or other forms of diabetes
* Patients with type 2 diabetes who are on no medications (diet-controlled), or metformin only unless they are within one year of diabetes onset
* Patients with significant cognitive, physical, or mental disability requiring that their diabetes care be managed by another individual (i.e. parent, spouse, guardian, nurse, residential facility) more than 25% of the time
* Non-English speaking
* Patients who are pregnant

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Visit completion rate in patients seen in the collaborative care and usual care models | 12 months
  Mean number of completed visits compared to scheduled visits (visit completion rate) in patients seen in the collaborative care and usual care models
Change in diabetes-related distress, measured by Problem Areas in Diabetes (PAID) | 12 months
  Problems Areas in Diabetes (PAID) is a validated screening tool for diabetes-related distress. Will measure change in PAID scores for both arms. The minimum score is 0 and maximum score is 80. The higher the score, the more severe diabetes-related distress.

SECONDARY OUTCOMES:
Change in HbA1c | 12 months
  Change in hemoglobin A1c
Change in mood, measured by Patient Health Questionnaire-8 (PHQ-8) | 12 months
  Patient Health Questionnaire-8 (PHQ-8) is a validated screening tool for depression. The minimum score is 0 and maximum score is 24. The higher the score, the more severe depression.
Change in anxiety, measured by Generalized Anxiety Disorder Scale-7(GAD-7) | 12 months
  Generalized Anxiety Disorder Scale-7(GAD-7) is a validated screening tool for anxiety. The minimum score is 0 and maximum score is 21. The higher the score, the more severe anxiety.
Change in Problem Areas in Diabetes (PAID) scores among those with score of 40 or higher at baseline, indicating moderate distress | 12 months
  Problems Areas in Diabetes (PAID) is a validated screening tool for diabetes-related distress. Will measure change in PAID scores for both arms. The minimum score is 0 and maximum score is 80. The higher the score, the more severe diabetes-related distress.
Change in disordered eating behavior, measured by Diabetes Eating Problem Survey- Revised (DEPS-R) | 12 months
  Diabetes Eating Problem Survey- Revised (DEPS-R) is a validated screening tool for disordered eating behavior for patients with diabetes on insulin therapy. The minimum score is 0 and maximum score is 75. The higher the score, the most severe disordered eating behavior.
Change in alcohol use, measured by Alcohol Use Disorders Identification Test Consumption (AUDIT-C) | 12 months
  Alcohol Use Disorders Identification Test Consumption (AUDIT-C) is a three-item self-administered screening test for alcohol misuse, validated in adults 18 years and older.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah J Wexler, MD, MSc, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Pilot and Feasibility study, no plan to share IPD